CLINICAL TRIAL: NCT00505050
Title: A Long-Term Prospective Randomized Controlled Study Using Repetitive Education at Six-Month Intervals and Monitoring for Adherence in Heart Failure Outpatients - The REMADHE Study
Acronym: REMADHE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 829/99
Record Dates: First submitted 2007-07-18; First posted 2007-07-20 (Estimated); Last update posted 2007-07-20 (Estimated); Status verified 2007-07

CONDITIONS: Heart Failure
Keywords: heart failure, disease program management, treatment, education
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (No Intervention): Standard follow-up medical visits and treatment for control group were performed during the study period by the same cardiologist team that was not informed of the randomization.
  Interventions: Other: Disease Program Management

INTERVENTIONS:
Other: Disease Program Management — This DMP inclused intervention content with education for out patients and caregivers; medication management with optimized therapy based on guidelines, and remote monitoring; delivery personnel with nurses, cardiologists, pharmacists, social workers, dietitians, physical therapists, psychologists; face-to-face individual/group communication, and telephone in-person; the intensity/complexity was long-term follow-up with 6 months interval repetitive education; the environment was hospital out-patient; and the outcomes measured were clinical, quality of life, and adherence.
  After randomization patients undergone our multidisciplinary education sessions 60-minute long that covered the basic principles related to heart failure. Telephone calls were used to reinforce the contents of the sessions of the ambulatory education activity, and monitoring of the compliance/adherence, symptoms/signs of worsening heart failure, and self-control mechanisms.

SUMMARY:
Recent meta-analysis reported reduction in mortality and hospitalization of HF patients.However, important issues in DMP for HF remain to be resolved. DMP are not homogeneous concerning methodology and in general included only elderly patients; most were tested in high-risk HF patients discharged from hospital; quality of life results are controversial; few reports included long-term results; some protocols had limited enrollment of screened patients, and it was suggested that could be less effective when patients are already followed by HF specialist.Improved survival was associated with cardiologist care as well with multidisciplinary teams providing specialized follow-up.Whether both together could benefits HF is not well defined. Also, no studies reported the long-term effects of a cyclic repetitive reeducation program.We tested whether a DMP that consisted of a long-term repetitive education program associated with a telephone monitoring could benefit HF outpatients in usual ambulatory care already under care of cardiologist with experience in HF

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients on ambulatory care were aged 18 years or older with irreversible chronic heart .failure with at least 6 months duration, and non planned surgical procedure or other procedure that could influence the follow-up in the next 6 months

Exclusion Criteria:

* impossibility for attendance of education sessions and monitoring based on non corrected limitations of transport, or unfavorable distance, or social, or of communication; myocardial infarction or unstable angina within 6 months before randomization; cardiac surgery or angioplasty within 6 months randomization; hospitalized patients or recent discharged patients; severe renal/hepatic/neurological/pulmonary or any systemic disease that could confuse the interpretation of results and impair expected survival; and pregnant women or women of childbearing potential.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-10; Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
The prespecified primary end-points were (1) combined death secondary to any cause or unplanned first hospitalization and (2) quality of life changes.

SECONDARY OUTCOMES:
(1) DMP feasibility;(2) death;(3)number and duration of hospitalization; (4) unexpected death in home and death during hospitalization; (5)emergency care necessity,(5) adherence.

CONTACTS AND LOCATIONS:
Overall Officials: Edimar Bocchi, Principal Investigator — Heart Institute of São University Medical School
Locations (1):
- Heart Institute of São Paulo University Medical School, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Ayub-Ferreira SM, Mangini S, Issa VS, Cruz FD, Bacal F, Guimaraes GV, Chizzola PR, Conceicao-Souza GE, Marcondes-Braga FG, Bocchi EA. Mode of death on Chagas heart disease: comparison with other etiologies. a subanalysis of the REMADHE prospective trial. PLoS Negl Trop Dis. 2013 Apr 25;7(4):e2176. doi: 10.1371/journal.pntd.0002176. Print 2013. PMID 23638197
- [Derived] Cruz Fd, Issa VS, Ayub-Ferreira SM, Chizzola PR, Souza GE, Moreira LF, Lanz-Luces JR, Bocchi EA. Effect of a sequential education and monitoring programme on quality-of-life components in heart failure. Eur J Heart Fail. 2010 Sep;12(9):1009-15. doi: 10.1093/eurjhf/hfq130. Epub 2010 Jul 29. PMID 20670963
- [Derived] Issa VS, Amaral AF, Cruz FD, Ayub-Ferreira SM, Guimaraes GV, Chizzola PR, Souza GE, Bocchi EA. Glycemia and prognosis of patients with chronic heart failure--subanalysis of the Long-term Prospective Randomized Controlled Study Using Repetitive Education at Six-Month Intervals and Monitoring for Adherence in Heart Failure Outpatients (REMADHE) trial. Am Heart J. 2010 Jan;159(1):90-7. doi: 10.1016/j.ahj.2009.10.027. PMID 20102872
- [Derived] Issa VS, Amaral AF, Cruz FD, Ferreira SM, Guimaraes GV, Chizzola PR, Souza GE, Bacal F, Bocchi EA. Beta-blocker therapy and mortality of patients with Chagas cardiomyopathy: a subanalysis of the REMADHE prospective trial. Circ Heart Fail. 2010 Jan;3(1):82-8. doi: 10.1161/CIRCHEARTFAILURE.109.882035. Epub 2009 Nov 20. PMID 19933408